CLINICAL TRIAL: NCT05391230
Title: IGHID 12128 - Getting Malaria "Off the Backs" of Women and Children in Western Uganda
Brief Title: Permethrin-treated Baby-wraps for the Prevention of Malaria in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-2569
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Malaria; P. Falciparum
Keywords: Permethrin; Plasmodium Falciparum Infection; Insecticide; Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized controlled trial of permethrin-treated lesus to prevent P. falciparum malaria in children 6-18 months of age. Study enrollment conducted at two sites in rural western Uganda. Participants will be randomized to one of two arms: permethrin-treated (intervention) or untreated (control) lesus. Participating mother-infant pairs will receive a new Long-lasting Insecticidal Net and two permethrin-treated or untreated lesus at enrollment. Total sample size will be 400 mother-infant pairs with 200 pairs in each arm. Participants will be followed longitudinally for six months, instructed and incentivized to present to one of the two study clinics when a fever develops, where they will be evaluated, tested, and treated, if positive, for malaria. Participants will attend scheduled clinic visits every two weeks for routine surveillance of adverse effects and tested for asymptomatic infection. Re-treatment and sham re-treatment of lesus will occur monthly.
Who Masked: Participant, Care Provider
Masking Description: Double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm : Arm that received permethrin-treated lesu (Experimental): Intervention Arm is the group that receives permethrin-treated lesu for use. The lesus of participants in the intervention group will be treated and subsequently retreated each month with 0.5% permethrin (Sawyer Products, Safety Harbor, FL).
  Interventions: Other: Permethrin-treated lesu
- Control Arm: Arm that received none permethrin-treated lesu (Sham Comparator): The lesus of participants in the control group will undergo sham treatment and re-treatment in which the cloth is soaked in water for a period of time similar to that of the intervention group. Participants and clinical staff (but not administrative staff) will be blinded to group assignments.
  Interventions: Other: Untreated lesu

INTERVENTIONS:
Other: Permethrin-treated lesu — 0.5% permethrin soaked baby wraps (lesus)
  Arms: Intervention Arm : Arm that received permethrin-treated lesu
Other: Untreated lesu — Water soaked baby wraps (lesus)
  Arms: Control Arm: Arm that received none permethrin-treated lesu

SUMMARY:
The scientific objective of this study is to test the protective effect of permethrin-treated lesus against P. falciparum malaria in infants and young children.

DETAILED DESCRIPTION:
General Study Design: The proposed study is a double-blind, randomized control trial of permethrin-treated lesus to prevent P. falciparum malaria in children 6-24 months of age conducted at two sites in rural western Uganda. Participating mother-infant pairs will receive a new bed net and two permethrin-treated or untreated lesus at enrollment. The total sample size will be 400 mother-infant pairs with 200 pairs in each group. The investigators will follow participants longitudinally for six months. Participants will be instructed and incentivized to present to one of the two study clinics when a fever develops, where they will be evaluated, tested, and treated, if positive, for malaria. Participants will also attend scheduled clinic visits every two weeks for routine surveillance of adverse effects and to test for asymptomatic infection. Re-treatment and sham re-treatment of lesus will occur each month.

Outcome Measures: The primary outcome measure is the incidence rate ratio of clinical (i.e., symptomatic) P. falciparum malaria in infants and children 6 - 24 months of age. Differences in malaria infection between treatment groups will be estimated with the incidence rate ratio, defined as the ratio of the number of clinical malaria episodes per 100 person-weeks at risk in the intervention group relative to the control group. This measure was chosen as it represents the most patient-centered measure of malaria burden, reflecting not only the potential negative health consequences, but also opportunity costs associated with care seeking and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form (ICF)
* Willing to comply with all study procedures and be available for the duration of the study
* Female of any age with a child 6 to 18 months of age at the time of enrollment
* Resident of village located in Bugoye, Maliba, or Mubuku sub-counties. Recruitment will initially focus on residents of villages within 2 km of study clinics in order to facilitate attendance, but we will not restrict enrollment to residents of these villages.

Exclusion Criteria:

* Mother or child taking any malaria chemoprevention regimen, including individuals living with HIV or exposed children who are taking cotrimoxazole that may modify risk of malaria
* Child with known sickle cell disease
* Known allergic reactions to components of the study product(s)
* Treatment with another investigational drug or other intervention
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female with infants between the ages of 6 months to 18 months at time of enrollment
Enrollment: 400 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-10-19 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical malaria in child | 7 days after onset of symptoms
  The presence of typical symptoms (e.g., fever, lethargy) and a positive malaria Rapid Diagnostic Test (RDT) during observation

SECONDARY OUTCOMES:
Change in child's hemoglobin level | (Week 0), Week 12, and Week 24 visits
  Change in child's hemoglobin as measured by HemoCue® device
Change in child's growth parameters | (Week 0), Week 12, and Week 24 visits
  Change in child's height and weight (e.g., weight and height will be combined to report BMI in kg/m^2).
Change in child's nutritional status | (Week 0), Week 12, and Week 24 visits using MUAC tape
  Change in child's mid-upper arm circumference (MUAC)
Prevalence of asymptomatic parasitemia | Every two weeks
  Presence of malaria parasites on bi-weekly dried blood spot (DBS) as determined by quantitative polymerase chain reaction(qPCR).
Malaria hospitalization | 14 days after onset of symptoms
  Child admitted to inpatient ward for treatment of malaria
Incidence of clinical malaria in mother | 7 days after onset of symptoms
  The presence of typical symptoms (e.g., fever, lethargy) and a positive malaria RDT during observation
Change in mother's hemoglobin level | (Week 0), Week 12, and Week 24 visits
  Change in child's hemoglobin as measured by HemoCue® device
Adverse reaction to permethrin treatment | 7 days after onset
  Self-reported history on bi-weekly questionnaire and confirmation by clinical staff.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Boyce, MD, Msc, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Mbarara University of Science and Technology (MUST), Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing through 36 months following publication
Access Criteria: Requesting investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Boyce RM, Shook-Sa BE, Ndizeye R, Baguma E, Giandomenico D, Cassidy CA, Eshun S, Siedner MJ, Staedke SG, Ntaro M, Juliano JJ, Reyes R, Mulogo EM. Permethrin-Treated Baby Wraps for the Prevention of Malaria. N Engl J Med. 2025 Oct 9;393(14):1399-1408. doi: 10.1056/NEJMoa2501628. Epub 2025 Sep 24. PMID 40991921
- [Derived] Boyce RM, Cassidy C, Ndizeye R, Baguma E, Giandomenico D, Shook-Sa BE, Ntaro M, Reyes R, Mulogo EM. Permethrin-treated baby wraps for the prevention of malaria in children: Protocol for a double-blind, randomized placebo-controlled controlled trial in western Uganda. PLoS One. 2023 Apr 27;18(4):e0284322. doi: 10.1371/journal.pone.0284322. eCollection 2023. PMID 37104305
- See also: Permethrin-treated baby wraps for the prevention of malaria: results of a randomized controlled pilot study in rural Uganda — https://malariajournal.biomedcentral.com/articles/10.1186/s12936-022-04086-w